CLINICAL TRIAL: NCT01437462
Title: Postoperative Pain After Propofol Sevoflurane Anaesthesia: a Prospective, Randomized, Single-blinded Trial
Brief Title: Sevoflurane, Propofol, Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Arvi Yli-Hankala, Professor, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Satu_Pokkinen_01_2011
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Healthy Adults; Gynecological Disease
Keywords: Pain, Postoperative; Anesthetics, intravenous; Anesthetics, inhalation; Otherwise healthy adults undergoing general anesthesia for gynecological disease.
MeSH Terms: conditions — Genital Diseases, Female; Pain, Postoperative; Respiratory Aspiration | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane inhalation anesthesia, sufficient amount to maintain adequate general anesthesia for surgery
  Other Names: Baxter Sevofluran
Drug: Propofol — Propofol intravenous anesthesia, sufficient amount to maintain adequate anesthesia during surgery
  Other Names: Propofol Lipuro

SUMMARY:
The impact of anaesthetic method (intravenous vs. inhalational) has been proposed, but not proven in a large-scale study. The researchers aim to provide an investigation that has sufficient power to clarify the potential effect of anaesthetic method on postoperative need of opioids. Sevoflurane and propofol will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years
* Gender: female
* ASA status 1-3
* Laparoscopic hysterectomy

Exclusion Criteria:

* Body Mass Index over 35
* Diabetes mellitus
* Liver disease
* Allergies to pharmaceuticals used in the Study
* Present use of opioids

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2008-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Postoperative consumption of an opioid (oxycodone) | 20 hours
  The consumption of oxycodone will be monitored by recording the amount of the drug received via a commercially available patient controlled analgesia (PCA) pump.

SECONDARY OUTCOMES:
NRS (numeral rating scale) of pain | 20 hours
  NRS is evaluated frequently during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Finland